CLINICAL TRIAL: NCT02770690
Title: the Effect of Ethyl Chloride Spray on Propofol Injection Pain
Brief Title: the Effect of Spray on Propofol Injection Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Young Eun Moon, Assistant Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CMC 2016-1
Record Dates: First submitted 2016-04-26; First posted 2016-05-12 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- spray (Experimental): apply the ethyl chloride spray before propofol injection
  Interventions: Drug: ethyl chloride spray
- lidocaine (Active Comparator): apply the lidocaine 0.5 mg/kg under the touniquette state before propofol injection
  Interventions: Drug: lidocaine
- placebo (Placebo Comparator): apply the saline before propofol injection
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ethyl chloride spray — apply the spray for 5 seconds on the dorsal hand before propofol iv injection
  Other Names: spray
  Arms: spray
Drug: lidocaine — apply lidocaine under the tourniquet state before propofol iv injection
  Arms: lidocaine
Drug: placebo — apply normal saline before propofol iv injection
  Other Names: normal saline
  Arms: placebo

SUMMARY:
While propofol is widely used an anesthetic induction medication, it causes the mild to moderate pain. Investigators will investigate the effect of ethyl chloride spray on propofol injection pain.

ELIGIBILITY:
Inclusion Criteria:

* the female patients undergoing hysteroscopy

Exclusion Criteria:

* the patients who are pregnant, have Raynaud's syndrome, or receive the pain killer

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
propofol injection pain | right after the propofol injection
  Propofol injection pain will be measured using the VAS (Visual analogue scale; 0cm=no pain, 10cm=the worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Youngeun Moon, MD, Principal Investigator — Assitant Professor
Locations (1):
- Youngeun Moon, Seoul, Seocho-gu, South Korea

IPD SHARING:
Plan to Share IPD: No